CLINICAL TRIAL: NCT01976780
Title: In Vivo and In Vitro Efficacy of Artemisinin Combination Therapy in Kisumu County, Western Kenya
Brief Title: In Vivo and In Vitro Efficacy of Artemisinin Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Global Emerging Infections Surveillance and Response System (U.S. Federal Agency)
Collaborators: United States Army Medical Unit - Kenya (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR1935
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Malaria
Keywords: Malaria; P. falciparum mono infection; Early Treatment Failure; Late Treatment Failure
MeSH Terms: conditions — Malaria | interventions — Artesunate; Artemether, Lumefantrine Drug Combination; Mefloquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS/MQ (Active Comparator): Treatment of P.falciparum mono-infection with 4 mg/kg of Artesunate daily for three days followed by 25mg/kg of Mefloquine split over two days.
  Interventions: Drug: Artesunate; Drug: Mefloquine
- AL (Active Comparator): Treatment of P. falciparum mono-infection with Artemether Lumefantrine administered at the standard dosage according to pre-defined weight bands (5-14 kg: 1 tablet; 15-24 kg: 2 tablets; 25-34 kg: 3 tablets; and > 34 kg: 4 tablets) given twice a day for 3 days.
  Interventions: Drug: Artemether Lumefantrine

INTERVENTIONS:
Drug: Artesunate
  Other Names: AS
  Arms: AS/MQ
Drug: Artemether Lumefantrine
  Other Names: AL
  Arms: AL
Drug: Mefloquine
  Other Names: MQ
  Arms: AS/MQ

SUMMARY:
This study aims to assess the degree of artemisinin resistance in adult and pediatric subjects presenting with uncomplicated falciparum malaria in Western Kenya. The study treatments will be Artemether Lumefantrine (AL) and Artesunate Mefloquine (ASMQ).

DETAILED DESCRIPTION:
Data generated by this study will provide a snapshot of the current situation regarding P. falciparum sensitivity to ACTs in Western Kenya. By having subjects in one of the study arms receive artesunate and then the partner drug after completion of the artemisinin phase will enable the accurate evaluation of the artemisinin derivative without the confounding influence of the partner drug. Sequential administration of the components of an ACT drug is recognized by the WHO as one of the ways in which ACTs can be administered. There will be close follow-up of the subjects throughout the duration of the study, and as such, subjects who fail to respond adequately will receive prompt rescue treatment. Since it is largely expected that most subjects in Western Kenya will have satisfactory responses to ACTs, data from this study will provide baseline information regarding parasite characteristics when compared to data from Thailand, an area that has reported resistance to ACTs. This, in turn, will potentially enable the identification of key markers, both in the host and the parasite, that may assist in the early detection of resistance, and also to better understand the development of resistance to ACTs. As such, the data generated from this study, both on its own and when compared to and pooled with data from similar studies that will be conducted in Peru and Thailand, will potentially inform both local and international policy regarding ACT use for the treatment of uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

* Adult/child aged between 6 months and 65 years inclusive (minimum weight 11kg), presenting with a measured temperature of ≥37.5 C, or history of fever within 24 hours prior to presentation
* Mono-infection with Plasmodium falciparum
* Baseline parasitemia of 2000 - 200,000 asexual parasites/µl
* Ability to provide informed consent
* Willingness and ability to comply with the study protocol for the duration of the study
* Willingness to remain in the hospital for 3 days

Exclusion Criteria:

* Presence of signs of severe malaria as defined by WHO
* Presence of severe anemia, defined as hemoglobin level below 6 g/dl
* Presence of mixed Plasmodium infection, or mono-infection of non-falciparum Plasmodium
* Inability to take oral medication
* History of allergy or contraindications to the study treatments
* Lactating or pregnant females
* Any condition that the investigator feels will result in an unfavorable outcome should the potential subject participate in the study

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Parasitological clearance rates by microscopy | 72 hours
  Clearance rates for the first 72 hour period after first ACT dose in patients with uncomplicated P. falciparum malaria

SECONDARY OUTCOMES:
Parasitological clearance rates by quantitative Polymerase Chain Reaction (PCR) | 72 hours
  PCR adjusted clearance rates for the first 72 hours after first ACT dose in patients with uncomplicated P. falciparum malaria
PCR-adjusted treatment efficacy of AL and AS/MQ | 42 days
Antimalarial drug sensitivity responses and molecular genotyping | 42 days
  Correlate clinical outcomes with results of above tests
Identify common specific genetic determinants of artemisinin resistance derived from parasite populations | 42 days
Gametocyte carriage in patients with uncomplicated malaria after treatment | 42 days
Catalog parasite samples | 42 days
  Correlated to clinical datasets to longitudinally track resistance trends
Pharmacokinetic parameters associated with ACT failure | 42 days

OTHER OUTCOMES:
Parasite clearance rates and immune response in semi-immune population | 42 days
  To assess the role of pre-existing semi-immunity against malaria in parasite clearance rates and immune response to acute infection
Production of microbiocidal molecules | 42 days
  To determine if stimulation of Peripheral Blood Mononuclear Cells (PBMC) (with MSP-1 or CSP antigens) elicit production of microbiocidal molecules (to be pursued only in if pre-existing immunity is shown to affect rate of clearance)
Acute cytokine response | 42 days
  To determine associations between the acute cytokine response with parasitemia clearance rates and immunologic responses

CONTACTS AND LOCATIONS:
Overall Officials: James F Cummings, MD, Study Chair — GEIS; Ben Andagalu, MD, Principal Investigator — Kenya Medical Research Institute/Walter Reed Project
Locations (1):
- Walter Reed Project, Kombewa Clinic, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Odhiambo G, Bergmann-Leitner E, Maraka M, Wanjala CNL, Duncan E, Waitumbi J, Andagalu B, Jura WGZO, Dutta S, Angov E, Ogutu BR, Kamau E, Ochiel D. Correlation Between Malaria-Specific Antibody Profiles and Responses to Artemisinin Combination Therapy for Treatment of Uncomplicated Malaria in Western Kenya. J Infect Dis. 2019 May 24;219(12):1969-1979. doi: 10.1093/infdis/jiz027. PMID 30649381